CLINICAL TRIAL: NCT01242241
Title: Propofol in Obese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Olutoyin A. Olutoye, Associate Professorof Anesthesiology & Pediatrics, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-22091
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Pharmacodynamics; Obesity
Keywords: Propofol; Childhood obesity; Pharmacodynamics
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-obese (Other): Non-obese children categorized as those with a body mass index(BMI)between 25-84th percentile
  Interventions: Drug: Propofol
- Obese children (Active Comparator): Obese children are categorized as those with a body mass index >95th percentile
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Each Obese child/subject in this group will receive a predetermined dose of propofol ranging from 1.0mg/kg to 4.25mg/kg to induce loss of consciousness depending on the response (presence or absence of lash reflex) of the preceding patient to his/her assigned dose (biased coin design)
  Other Names: Diprivan
  Arms: Obese children
Drug: Propofol — This arm of patients(non-obese)will act as the control group for the obese children. Each non-obese child/subject will receive a predetermined dose of propofol from a range of 1.0mg/kg to 4.25mg/kg depending on the response of the previous patient to their assigned dose( biased coin design)
  Other Names: Diprivan
  Arms: Non-obese

SUMMARY:
Obesity in children,as in adults,has rapidly become a public health concern. Studies in adults have shown that obesity, now considered to be a disease state, is a modifier of the effect of drugs on the body as well as how the body handles the drug.The anesthetic management of obese children poses a variety of significant challenges which include determination of the appropriate dose of anesthetic intravenous agents. Dosing of most drugs is calculated based on the effective dose in 50% of patients but the more practical and required information is the effective dose in 95%(ED95%)of patients. The aim of this study is to determine the effective dose in 95% of patients(children). The hypothesis is the ED95 of propofol in obese children will be higher than that of non-obese children.

DETAILED DESCRIPTION:
All subjects were fasted in keeping with our institutional NPO guidelines and had IV access established in the upper extremity in the pre-anesthesia area. No pre-induction sedative drugs were administered. Routine ASA monitors were applied and in cooperative children, a bispectral index (BIS) monitor pad (Aspect Medical Systems, Inc., Shattuck, MA) was applied over the forehead. Each child was given a water-filled syringe to hold tightly in the hand contralateral to the IV site. Lidocaine 1 mg/kg IV (maximum of 60 mg) was administered to decrease pain with propofol injection. A predetermined sequential dose of propofol (Diprivan, APP Pharmaceuticals, LLC, Schaumburg, IL) was administered IV rapidly over 10 seconds, followed by a normal saline flush.

Biased Coin Design An independent observer blinded to the propofol dose tested for lash reflex at 20 seconds, and also recorded the vital signs; level of sedation, using the University of Michigan sedation scale (UMSS)10; and the BIS values at 20, 60, and 120 seconds after propofol administration, along with the time the patient dropped the handheld syringe. The study was terminated after 120 seconds and additional propofol administered if needed.

Both nonobese and obese patients were studied in parallel using the biased coin design (BCD), in which a certain number of dose levels (k levels) are chosen with a fixed constant interval. In the absence of dose-ranging data in obese children, we chose a low starting dose of 1.0 mg/kg for the first patient in both groups to avoid missing a desired response in this patient population. If the desired effect (loss of lash reflex at 20 seconds) was not observed, the next patient in the assigned group received the next higher dose of propofol in predetermined increments (0.25 mg/kg) from the previous dose. If the desired effect was observed, the next patient in the same assigned group was randomized with a 0.95 probability to receive the same dose or a 0.05 probability to receive the next lower dose (also in 0.25 mg/kg decrements).

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 3 and 17 years who fall into the categories of non-obese(BMI percentile between 25-84th percentile) or obese(>95th percentile)
2. American Society of Anesthesiology(ASA) classification 1 or 2-

Exclusion Criteria:

1. Patients classified as ASA (American Society of Anesthesiology) Class 3 or greater.
2. Patients with documented kidney or liver disease or those presenting for open surgery on the liver or kidney.
3. Patients who will NOT be receiving propofol for induction as part of their anesthetic regimen.
4. Patients who are currently on anti-convulsant medication or receiving drugs with sedative effects.
5. Patients currently being treated for attention deficit disorder.
6. Patients who are diagnosed with failure to thrive or those with a BMI less than 25th percentile.
7. Patients who are hemodynamically unstable.
8. Patients with egg allergy.
9. Patients with low levels of albumin -

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olutoyin A Olutoye, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Mulla H, Johnson TN. Dosing dilemmas in obese children. Arch Dis Child Educ Pract Ed. 2010 Aug;95(4):112-7. doi: 10.1136/adc.2009.163055. Epub 2010 Jun 28. PMID 20585055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the operating room setting between the period of April 2008 to December 2011
Pre-assignment Details: A total of 213 patients were screened for study eligibility. Eighty-two patients were excluded; 51 did not meet inclusion criteria either becasue they declined participation, did not have intravenous access, were re-scheduled due to inadequate preparation for surgery or patient illness. All patients enrolled completed the study.
Groups:
- Obese Children: Obese children are categorized as those with a body mass index >95th percentile
  Propofol : Each Obese child/subject in this group received a predetermined dose of propofol ranging from 1.0mg/kg to 4.25mg/kg to induce loss of consciousness depending on the response (presence or absence of lash reflex) of the preceding patient to his/her assigned dose (biased coin design)
- Non-obese: Non-obese children categorized as those with a body mass index(BMI)between 25-84th percentile
  Propofol : This arm of patients(non-obese)served as the control group for the obese children. Each non-obese child/subject received a predetermined dose of propofol from a range of 1.0mg/kg to 4.25mg/kg depending on the response of the previous patient to their assigned dose( biased coin design)
Period: Overall Study
Arm/Group | Obese Children | Non-obese
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Children | Non-obese | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 40 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.69 (2.89) | 12.70 (3.90) | 12.69 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 22 | 24 | 46
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.29 (5.12) | 19.01 (2.60) | 24.65 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Dose of Propofol That Caused Loss of Consciousness in 95% (ED95) of Obese and Non-obese Children
Description: Propofol is administered over 10 seconds. 20 seconds after adminstration, loss of consciousness is assessed by the presence or absence of a lash reflex. The dose responsible for loss of lash reflex/consciousness in 95% of patients was determined in mg/kg.
Time Frame: 20 seconds
Population: The sample size of 40 patients in each group was based on previous simulation studies which used the biased coin design in which a group size of 20-40 patients was shown to demonstrate stable estimates of the target dose for most scenarios.
Measure: Median (Full Range); unit: mg/kg
Arm/Group | Obese Children | Non-obese
Number analyzed (Participants) | 40 | 40
mg/kg | 2 [1 to 2.25] | 2.125 [1 to 3.25]

2. Secondary Outcome: Depth of Sedation
Description: After propofol administration, the patient was assessed for depth of sedation at 30 seconds, 1 minute, and 2 minutes using the University of Michigan Sedation Scale (UMSS) and Ramsay Sedation Scale. UMSS assesses the level of alertness on a five-point scale ranging from 1 (wide awake) to 5 (unarousable with deep stimulation). Ramsay Sedation Scale assesses the level of sedation on a six-point scale ranging from 1 (Patient is anxious and agitated or restless, or both) to 6 (Patient exhibits no response).
Time Frame: 30 seconds, 1 minute, and 2 minutes
Population: Due to unavoidable circumstances during a clinical surgery, depth of sedation was not able to be collected on every subject at every time point.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Obese Children | Non-obese
Number analyzed (Participants) | 40 | 40
units on a scale
  UMSS - 30 seconds: number analyzed (Participants) | 37 | 37
  UMSS - 30 seconds | 3.65 [1 to 4] | 3.57 [1 to 4]
  UMSS - 1 minute: number analyzed (Participants) | 37 | 37
  UMSS - 1 minute | 3.86 [1 to 4] | 3.73 [1 to 4]
  UMSS - 2 minutes: number analyzed (Participants) | 38 | 39
  UMSS - 2 minutes | 3.82 [1 to 4] | 3.67 [1 to 4]
  Ramsay - 30 seconds: number analyzed (Participants) | 35 | 34
  Ramsay - 30 seconds | 5.74 [2 to 6] | 5.71 [1 to 6]
  Ramsay - 1 minute: number analyzed (Participants) | 37 | 35
  Ramsay - 1 minute | 5.92 [4 to 6] | 5.83 [2 to 6]
  Ramsay - 2 minutes: number analyzed (Participants) | 37 | 35
  Ramsay - 2 minutes | 5.92 [4 to 6] | 5.86 [2 to 6]

ADVERSE EVENTS:
Time Frame: From 0-120 seconds of propofol administration
Arm/Group | Non-obese | Obese Children
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT01242241/Prot_SAP_000.pdf